CLINICAL TRIAL: NCT06679816
Title: Study on the Efficacy of Hydrocortisone in Perioperative Hormone Replacement Therapy for Large Pituitary Neuroendocrine Tumors:a Multicenter, Randomized, Double-blind, Placebo- Parallel Controlled Study
Brief Title: Hydrocortisone in Hormone Replacement Therapy for Large Pituitary Neuroendocrine Tumors
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HEALTH
Record Dates: First submitted 2024-11-06; First posted 2024-11-08 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-12

CONDITIONS: Pituitary Adenoma; Pituitary Neuroendocrine Tumor
MeSH Terms: conditions — Pituitary Neoplasms | interventions — Hormone Replacement Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hormone supplementation therapy group (Experimental)
  Interventions: Drug: Hormone replacement therapy
- Placebo therapy group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hormone replacement therapy — Perioperative Hydrocortisone Reduction Therapy
  Arms: Hormone supplementation therapy group
Drug: Placebo — Perioperative placebo Reduction Therapy
  Arms: Placebo therapy group

SUMMARY:
The goal of this clinical trial is to assess the need for hydrocortisone replacement therapy during the perioperative period for large pituitary neuroendocrine tumors. The main questions it aims to answer are:

• Does hydrocortisone replacement therapy reduce the incidence of adrenal insufficiency in participants? Researchers will compare hydrocortisone to a placebo (a look-alike substance that contains no drug) to see if hydrocortisone works to reduce the incidence of adrenal insufficiency.

Participants will:

* Take or intravenous infusion drug hydrocortisone or a placebo every day for 2 weeks
* Visit the clinic three months after surgery for checkups and tests
* Keep a diary of their symptoms

ELIGIBILITY:
Inclusion Criteria:

* (1) Age range: 18-70 years old;
* (2) Accept PitNETs patients who can be treated with endoscopic transsphenoidal surgery;
* (3) The maximum diameter of the tumor is ≥ 2 centimeters;
* (4) Preoperative hypothalamic pituitary adrenal axis integrity;
* (5) The subject or their legal representative signs the informed consent form

Exclusion Criteria:

* (1) Patients with a history of Cushing's disease or adrenal insufficiency;
* (2) Emergency and combined hormone therapy patients;
* (3) Pituitary stroke patients;
* (4) Patients lacking head magnetic resonance imaging;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 882 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of adrenal insufficiency on the first or second day after surgery | the first or second day after surgery

SECONDARY OUTCOMES:
The incidence of adrenal insufficiency within 90 days after surgery | Within 90 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing, Beijing Tiantan Hospital,Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Research data involves subject privacy